CLINICAL TRIAL: NCT06483178
Title: A Randomised Controlled Trial Comparing Gait in Fixed or Rotating Cementless Total Knee Arthroplasties
Brief Title: Gait in Fixed Or Rotating Cementless Total Knee Arthroplasties
Acronym: G-FORCE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: Imperial College London (Other); Trauma and Orthopaedics Research Charity (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21057RN-SW
Record Dates: First submitted 2024-01-31; First posted 2024-07-03 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Total Knee Arthroplasty; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: A single centred, parallel group, randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Attune (Experimental)
  Interventions: Device: Attune knee implant
- Triathlon (Active Comparator)
  Interventions: Device: Triathlon knee implant

INTERVENTIONS:
Device: Attune knee implant — Attune cementless cruciate retaining rotating platform implant (DePuy Synthes) with a standard gap balancing cruciate sacrificing surgical technique
  Arms: Attune
Device: Triathlon knee implant — Triathlon cementless condylar stabilised implant (Stryker) with a standard gap balancing cruciate sacrificing surgical technique
  Arms: Triathlon

SUMMARY:
The number of patients requiring knee replacements is increasing every year due to the combination of an aging population, increased patient expectancy, and rising levels of obesity. Therefore, newer implants, or design features, are introduced on a regular basis to try to improve patient outcomes. In 2013, DePuy Synthes launched the Attune Knee System to provide improved range of motion and address the unstable feeling some patients experience whilst performing everyday activities, such as going down stairs. The Attune cementless rotating platform knee was first implanted in September 2016. In 2004, the first Triathlon total knee designed by Stryker was implanted. Registry figures for both the Attune and Triathlon knees are promising with good implant longevity and outcomes.

There is only a small amount of literature available on the Attune knee as it is still a relatively new implant. Worldwide, the Triathlon is widely used and is also a well-established, successful implant used in the investigators' unit. This study will help to determine whether the Attune can improve patient outcomes in terms of gait analysis assessed by walking on a treadmill, patient reported outcome measures and X-ray outcomes when compared to the Triathlon knee. 90 patients who will undergo knee replacement and meet the inclusion criteria and agree to take part will be randomly placed in one of two groups to receive either the Attune or Triathlon knee implant.

DETAILED DESCRIPTION:
The number of patients requiring Total Knee Arthroplasty (TKA) is increasing every year due to the combination of an aging population, increased patient expectancy, and rising levels of obesity which accelerates the onset of osteoarthritis. Therefore, newer implants, or design features, are introduced on a regular basis in an attempt to incrementally improve patient outcomes. In 2013, DePuy Synthes launched the Attune Knee System to provide improved range of motion (ROM) and address the unstable feeling some patients experience whilst performing everyday activities, such as descending stairs. The Attune Knee System features a gradually reducing femoral radius, an innovative s-curve design of the posteriorly stabilised cam, a tibial base which can be downsized or upsized two sizes versus the insert, novel patella tracking, lighter innovative instruments, and a new polyethylene formulation. These implant properties could potentially produce improved gait and speed, better stability of the knee in deep flexion, reduced joint forces, better patella tracking, improved operative flexibility and efficiency, and implant longevity. The system currently comprises 14 femoral sizes, 10 tibial sizes and 5 patella options.

Registry figures regarding the Attune Knee System are promising. The 2020 figures from the National Joint Registry (NJR) for England, Wales, Northern Ireland and the Isle of Man, show that the cumulative revision rate for the Attune knee (fixed bearing) was 2.7% (95% confidence interval (CI), 2.32-3.17) at 5 years (i.e. implant survivorship at 5 years of 97.3%) out of 25,723 knee joints. The cumulative revision rate for the Attune knee (rotating platform (RP)) was 1.7% (95% CI, 1.17-2.50) at 5 years (i.e. implant survivorship at 5 years of 98.3%) out of 4,254 knee joints. Figures from the Australian Orthopaedic Association National Joint Replacement Registry (AOANJRR) 2020 Report show that the 5-year cumulative revision rate of the Attune Cruciate Retaining implant was 3.0% (95% CI, 2.7 to 3.5) out of 15,300 knees. The 5-year cumulative revision rate of the Attune Posterior Stabilized (PS) implant was 2.6% (95% CI, 2.1 to 3.3) out of 7,179 knees.

The Attune cementless Rotating Platform was first implanted in September 2016 and by February of 2021 over 22,000 have been implanted worldwide. There are only a small number of studies regarding the Attune implant due to its infancy. In 2004, the first Triathlon total knee (Stryker) was implanted. The Triathlon knee was designed to address the main reasons for revision surgery such as instability, patellofemoral tracking complications and loosening/osteolysis. There are cruciate-retaining, condylar-stabilising, posterior-stabilising and difficult primary options available. The single radius design allows for mid-flexion stability. Over 3 million Triathlon knees have been implanted worldwide.

Joint registries show a high rate of survivorship of the Triathlon with over 10 years of follow up. The 2020 figures from the NJR for England, Wales, Northern Ireland and the Isle of Man, show that the cumulative revision rate for the Triathlon was 2.2% (95% CI, 2.10-2.20) at 5 years (i.e. implant survivorship at 5 years of 97.8%) and 3.4% (95% CI, 3.18-3.56) at 10 years (i.e. implant survivorship at 10 years of 96.6%) out of 133,729 knee joints. Figures from the AOANJRR 2020 Report show that the cumulative revision rate of the Triathlon CR implant was 2.5% (95% CI, 2.4 to 2.7) at 5 years and 3.9% (95% CI, 3.7 to 4.2) at 10 years out of a total 50,402 knees. The cumulative revision rate of the Triathlon PS implant was 4.0% (95% CI, 3.6 to 4.5) at 5 years and 6.1% (95% CI, 5.5 to 6.9) at 10 years out of a total 8,755 knees.

To the investigators' knowledge, the only study to compare the Attune and Triathlon TKAs was a retrospective cohort analysis in 2018 using cemented components. The Attune implant was received by 1,178 patients, whilst the Triathlon implant was received by 5,707 patients. Patients who received the Attune TKA had a statistically significantly shorter length of stay and operating room time, were statistically significantly less likely to be discharged to a skilled nursing facility or other inpatient facility, and had statistically significantly lower total hospital cost than those who received the Triathlon implant.

To date, the large majority of studies comparing the Attune TKA to other implants have used the PFC Sigma TKA as a comparator. Most of these studies have examined cemented implants only. A retrospective review comparing 114 PFC Sigma cemented and 103 Attune cemented TKAs with a mean follow-up of 3.2 years found similar rates of patellar crepitus clunk and anterior knee pain. There were also no clinically significant differences in ROM, pain, or Knee Society Score (KSS) between the two groups. Another retrospective review compared migration of the cemented Attune fixed bearing CR tibial component with the cemented PFC-sigma fixed bearing CR tibial component. The overall migration at two years of both groups (38 Attune and 36 PFC Sigma) was comparable: mean 1.13 mm (95% CI, 0.97 to 1.30) for the Attune and 1.16 mm (95% CI, 0.99 to 1.35) for the PFC-sigma. At two years, the mean backward tilting was -0.43° (95% CI, -0.65 to -0.21) for the Attune and 0.08° (95% CI -0.16 to 0.31) for the PFC-sigma. The clinical outcomes and Patient Reported Outcome Measures (PROMs) (Knee injury and Osteoarthritis Outcome Score (KOOS), pain scores, KSS and Oxford Knee Score (OKS)) improved between pre-operation and two years post-operation and were not significantly different between groups. Radiolucent lines (RLLs) at the implant-cement interface were mainly seen below the medial tibial baseplate in 17% of the Attune patients and 3% of the PFC-sigma patients at two weeks (no significant difference), and at two years 42% and 9% of patients respectively (p=0.001). All implant-cement interface radiolucencies were less than 2 mm. It was noted that the version of the Attune tibial component examined in this study had since undergone modification by the manufacturer. In a further randomised controlled trial of 80 cemented Attune and 78 cemented PFC Sigma TKAs, there were no significant differences found in post-operative KSS, Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), ROM or Visual Analogue Scale (VAS) pain score between the two groups at 2-year follow-up. Both groups showed significantly improved outcomes 2 years after surgery.

Thirty TKA patients (15 Attune and 15 Sigma both CR FB) with a KOOS>70 and at least 1 year post-operation were assessed during five complete cycles of level walking, stair descent (0.18-m steps), deep knee bend, and sitting down onto and standing up from a chair, using a moving fluoroscope (25 Hz, 1 ms shutter time). Kinematic data were extracted by 2D/3D image registration. The results demonstrated similar tibiofemoral ranges of motion for flexion-extension, abduction-adduction, internal-external rotation, and anteroposterior (AP) translation for both groups. The pattern of AP translation-flexion-coupling differed between the two groups. The subjects with the Sigma TKA showed a sudden change in direction of AP translation around 30º of flexion, which was not present in the subjects with the Attune patients.

Musgrave Park Hospital (MPH) is one of the largest Orthopaedic centres in the United Kingdom (UK) performing more than 1,000 primary TKAs annually. It is part of the Belfast Health and Social Care Trust (BHSCT) in Northern Ireland. Nearly 1,000 Attune TKAs have been performed in MPH since 2022, with over 1,000 cementless Triathlons in more recent years.

MPH has a Compact Tandem Force-Sensing Treadmill (DBCEEWI-CE, AMTI Force and Motion, Watertown, MA, USA) capable of measuring vertical, anteroposterior and mediolateral forces and moments. It can measure 6 ground reaction force components (Fx,Fy,Fz, Mx,My,Mz), with a variable speed of 0-18 Km/h, linearity of <±0.5% full scale output, hysteresis of <±0.5% full scale output and maximum inclination 25% grade. This study will be in collaboration with Professor Justin Cobb's research team in Imperial College, London who have established expertise in this form of gait analysis. The Total or Partial Knee Arthroplasty Trial (TOPKAT) randomised controlled trial which included 264 total and 264 partial knees reported no significant differences in OKS between the two groups. At MPH, a subgroup of these patients (16 total knees, 11 partial knees and 16 volunteers with no knee replacements) completed post-operative gait analysis at a mean of 4.5 years following surgery. Analysis of this data showed no differences in gait symmetry between the two groups during level, downhill and uphill walking. Both groups demonstrated similar gait profiles during the three walking conditions to that of the healthy volunteers.

Design features of Attune vs Triathlon There are two key design features which are different between the Attune and Triathlon TKAs.

1. Coronal stability due to sagittal kinematics design. The Attune knee has a Gradually-Reducing radius of curvature termed the Attune Gradius curve from 5-65º flexion. The Triathlon has a Single Radius design from 10-110º flexion.
2. Sagittal (AP stability) variation due to Triathlon's 'Rotatory Arc' which attempts to achieve some rotational freedom to compensate for the Single Radius design but comes at the expense of increased AP laxity.

Rationale for the Study: To date, there has been a paucity of literature on the Attune TKA as it is still a relatively new implant. Worldwide, the Triathlon is widely used and is also a well-established, successful implant used in the investigators' unit. The single radius of the Triathlon may provide a less stable knee joint compared to the gradually reducing curve of the Attune knee which provides AP stability and greater ROM. The Triathlon TKA has approximately 5.6 mm of AP laxity but the literature suggests >10 mm of AP laxity is associated with a reduction in functional outcome scores. Therefore, the primary outcome of gait analysis is being used in this study as a more sensitive measure of knee function. Both the Attune and Triathlon TKAs have been designed with a similar evolution of the trochlear geometry - both are asymmetric laterally. This study will be able to determine whether the Attune can improve patient outcomes in terms of gait analysis, patient reported outcome measures and radiological outcomes. Based on previous work from Professor Justin Cobb's research team in Imperial College, London, it is postulated that gait analysis assessed on a decline will demonstrate a difference between the aforementioned Attune and Triathlon design philosophies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged <65 years old who require a primary TKA for medial compartment osteoarthritis with a varus deformity.
* On examination patients must have a pain free ROM of both hips, both ankles and the opposite knee. A history of mild pain in any of these lower limb joints that does not inhibit mobility is acceptable.
* Must be able to walk at a pre-operative speed of at least 4 km/h (approximately 30 metres in 30 seconds).
* Must be able to walk outside unaided or with no more than a walking stick.
* Must be able to complete pre- and post-operative gait analysis.
* Participants must have a functional level of spoken and written English and must have a smartphone or have access to a smartphone to complete the online questionnaires on REDCap and to take photographs for virtual assessment of ROM.

Exclusion Criteria:

* Patients with valgus deformity of the knee.
* Patients with previous lower limb arthroplasty.
* Patients with previous lower limb open reduction and internal fixation (ORIF).
* Patients who are American Society of Anaesthesiologists (ASA) grade 3 or higher.
* Patients who are unable to adhere to the trial protocol (due to cognitive impairment, cannot speak English or for any other reason).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Post-operative top downhill walking speed at 9-12 months. | 9-12 months
  Post-operative top downhill walking speed at 9-12 months will be assessed via gait analysis.

SECONDARY OUTCOMES:
Ground reaction forces in the vertical plane throughout the stance phase of the gait cycle. | 9-12 months
Ground reaction forces in the medio lateral plane throughout the stance phase of the gait cycle. | 9-12 months
Ground reaction forces in the anterior posterior plane throughout the stance phase of the gait cycle. | 9-12 months
Gait symmetry at weight acceptance (heel strike) of the stance phase | 9-12 months
Gait symmetry at mid-stance of the stance phase | 9-12 months
Gait symmetry at push off of the stance phase | 9-12 months
Spatiotemporal gait parameter - step length | 9-12 months
Spatiotemporal gait parameter - stride length | 9-12 months
Spatiotemporal gait parameter - step width | 9-12 months
Spatiotemporal gait parameter - step time | 9-12 months
Spatiotemporal gait parameter - double support time | 9-12 months
Pain Visual Analogue Score (VAS) | Pre-operation, post-operatively weekly from Week 1 to Week 6, 3 months and 12 months.
  The Pain VAS score will be completed by participants online with a score ranging from zero to 100 with 0 being no pain and 100 being worst pain imaginable.
Oxford Knee Score (OKS) | Pre-operation, 3 months and 12 months.
  The OKS will be completed by participants online, with a score ranging from 0 (worst score possible) - 48 (best score possible).
EuroQoL-5D (EQ-5D-5L) | Pre-operation, 3 months and 12 months.
  The EQ-5D-5L will be completed by participants online. A single score will be derived which ranges from -0.594 to 1, where 0 is death and 1 is full health.
EuroQoL-5D Visual Analogue Scale (VAS) | Pre-operation, 3 months and 12 months.
  The EQ-5D VAS will also be scored from 0 (worst health possible) - 100 (best health possible).
Forgotten Joint Score (FJS) | Pre-operation, 3 months and 12 months.
  The FJS will also be completed by participants online, with every question scored 1 (never) to 5 (mostly). The raw score ranges from 12 to 60 and this score is then used to give a final score with the higher the score the better outcome.
  Final score = 100 - ((sum (Item 1 to Item 12) - 12)/48*100)
Feller's Patellar score | Pre-operation, 3 months and 12 months.
  The questionnaire includes items on anterior knee pain, quadriceps strength, ability to rise from a chair and climb stairs; these scores range from 3 to 30 points, with 30 points representing the best possible score.
Range of motion (ROM) | Pre-operation, 6 weeks, 3 months and 12 months.
  ROM will be assessed face-to-face pre-operatively, virtually at 6 weeks, and face-to-face at 3 months and 12 months if convenient for the patient. If ROM cannot be taken face-to-face at 3 months or 12 months, ROM will be assessed virtually. To do this, participants will email photos of their knee following guidance from a participant information sheet. These photos will then be uploaded to the DrGoniometer app to take the measurements of ROM. Three readings of ROM will be recorded:
  1. Extension
  2. Active flexion
  3. Forced passive flexion performed by the participant
Length of stay in hospital | Up to 4 months
  Total length of stay in hospital will be calculated using date of discharge and date of operation.
90-day complications | 3 months
  This will include Out of Hour attendances, A&E attendances, readmissions to hospital and any returns to theatre.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Napier, Principal Investigator — Belfast Health and Social Care Trust
Locations (1):
- Musgrave Park Hospital, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carey BW, Harty J. A comparison of clinical- and patient-reported outcomes of the cemented ATTUNE and PFC sigma fixed bearing cruciate sacrificing knee systems in patients who underwent total knee replacement with both prostheses in opposite knees. J Orthop Surg Res. 2018 Mar 15;13(1):54. doi: 10.1186/s13018-018-0757-6. PMID 29544516
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Bonutti PM, Khlopas A, Chughtai M, Cole C, Gwam CU, Harwin SF, Whited B, Omiyi DE, Drumm JE. Unusually High Rate of Early Failure of Tibial Component in ATTUNE Total Knee Arthroplasty System at Implant-Cement Interface. J Knee Surg. 2017 Jun;30(5):435-439. doi: 10.1055/s-0037-1603756. Epub 2017 Jun 7. No abstract available. PMID 28591930
- [Background] Indelli PF, Pipino G, Johnson P, Graceffa A, Marcucci M. Posterior-stabilized total knee arthroplasty: a matched pair analysis of a classic and its evolutional design. Arthroplast Today. 2016 Aug 21;2(4):193-198. doi: 10.1016/j.artd.2016.05.002. eCollection 2016 Dec. PMID 28326427
- [Background] Etter K, Lerner J, Kalsekar I, de Moor C, Yoo A, Swank M. Comparative Analysis of Hospital Length of Stay and Discharge Status of Two Contemporary Primary Total Knee Systems. J Knee Surg. 2018 Jul;31(6):541-550. doi: 10.1055/s-0037-1604442. Epub 2017 Aug 25. PMID 28841727
- [Background] Bateman DK, Preston JS, Mennona S, Gui E, Kayiaros S. Comparison Between the Attune and PFC Sigma in Total Knee Arthroplasty: No Difference in Patellar Clunk and Crepitus or Anterior Knee Pain. Orthopedics. 2020 Nov 1;43(6):e508-e514. doi: 10.3928/01477447-20200812-05. Epub 2020 Aug 20. PMID 32818287
- [Background] Kaptein BL, den Hollander P, Thomassen B, Fiocco M, Nelissen RGHH. A randomized controlled trial comparing tibial migration of the ATTUNE cemented cruciate-retaining knee prosthesis with the PFC-sigma design. Bone Joint J. 2020 Sep;102-B(9):1158-1166. doi: 10.1302/0301-620X.102B9.BJJ-2020-0096.R1. PMID 32862688
- [Background] Hauer G, Horlesberger N, Klim S, Bernhardt GA, Leitner L, Glehr M, Leithner A, Sadoghi P. Mid-term results show no significant difference in postoperative clinical outcome, pain and range of motion between a well-established total knee arthroplasty design and its successor: a prospective, randomized, controlled trial. Knee Surg Sports Traumatol Arthrosc. 2021 Mar;29(3):827-831. doi: 10.1007/s00167-020-06027-z. Epub 2020 Apr 24. PMID 32333057
- [Background] Hamilton WG, Brenkel IJ, Barnett SL, Allen PW, Dwyer KA, Lesko JP, Kantor SR, Clatworthy MG. Comparison of Existing and New Total Knee Arthroplasty Implant Systems From the Same Manufacturer: A Prospective, Multicenter Study. J Am Acad Orthop Surg Glob Res Rev. 2021 Dec 15;5(12):e21.00136. doi: 10.5435/JAAOSGlobal-D-21-00136. PMID 34908561
- [Background] Molloy IB, Keeney BJ, Sparks MB, Paddock NG, Koenig KM, Moschetti WE, Jevsevar DS. Short term patient outcomes after total knee arthroplasty: Does the implant matter? Knee. 2019 Jun;26(3):687-699. doi: 10.1016/j.knee.2019.01.018. Epub 2019 Mar 23. PMID 30910627
- [Background] Chua JL, Goh GS, Liow MHL, Tay DK, Lo NN, Yeo SJ. Modern TKA implants are equivalent to traditional TKA implants in functional and patellofemoral joint-related outcomes. Knee Surg Sports Traumatol Arthrosc. 2019 Apr;27(4):1116-1123. doi: 10.1007/s00167-018-5161-6. Epub 2018 Sep 29. PMID 30269170
- [Background] Staats K, Wannmacher T, Weihs V, Koller U, Kubista B, Windhager R. Modern cemented total knee arthroplasty design shows a higher incidence of radiolucent lines compared to its predecessor. Knee Surg Sports Traumatol Arthrosc. 2019 Apr;27(4):1148-1155. doi: 10.1007/s00167-018-5130-0. Epub 2018 Sep 22. PMID 30244340
- [Background] Ranawat CS, White PB, West S, Ranawat AS. Clinical and Radiographic Results of Attune and PFC Sigma Knee Designs at 2-Year Follow-Up: A Prospective Matched-Pair Analysis. J Arthroplasty. 2017 Feb;32(2):431-436. doi: 10.1016/j.arth.2016.07.021. Epub 2016 Aug 9. PMID 27600300
- [Background] Song SJ, Park CH, Liang H, Kang SG, Park JJ, Bae DK. Comparison of Clinical Results and Injury Risk of Posterior Tibial Cortex Between Attune and Press Fit Condylar Sigma Knee Systems. J Arthroplasty. 2018 Feb;33(2):391-397. doi: 10.1016/j.arth.2017.09.056. Epub 2017 Oct 6. PMID 29066248
- [Background] Saffarini M, Demey G, Nover L, Dejour D. Evolution of trochlear compartment geometry in total knee arthroplasty. Ann Transl Med. 2016 Jan;4(1):7. doi: 10.3978/j.issn.2305-5839.2015.12.53. PMID 26855943
- [Background] Webb JE, Yang HY, Collins JE, Losina E, Thornhill TS, Katz JN. The Evolution of Implant Design Decreases the Incidence of Lateral Release in Primary Total Knee Arthroplasty. J Arthroplasty. 2017 May;32(5):1505-1509. doi: 10.1016/j.arth.2016.11.050. Epub 2016 Dec 14. PMID 28089467
- [Background] Martin JR, Jennings JM, Watters TS, Levy DL, McNabb DC, Dennis DA. Femoral Implant Design Modification Decreases the Incidence of Patellar Crepitus in Total Knee Arthroplasty. J Arthroplasty. 2017 Apr;32(4):1310-1313. doi: 10.1016/j.arth.2016.11.025. Epub 2016 Nov 22. PMID 28012722
- [Background] Toomey SD, Daccach JA, Shah JC, Himden SE, Lesko JP, Hamilton WG. Comparative Incidence of Patellofemoral Complications Between 2 Total Knee Arthroplasty Systems in a Multicenter, Prospective Clinical Study. J Arthroplasty. 2017 Sep;32(9S):S187-S192. doi: 10.1016/j.arth.2017.04.014. Epub 2017 Apr 20. PMID 28600108
- [Background] Berahmani S, Hendriks M, Wolfson D, Wright A, Janssen D, Verdonschot N. Experimental pre-clinical assessment of the primary stability of two cementless femoral knee components. J Mech Behav Biomed Mater. 2017 Nov;75:322-329. doi: 10.1016/j.jmbbm.2017.07.043. Epub 2017 Jul 27. PMID 28779696
- [Background] Behrend H, Zdravkovic V, Bosch M, Hochreiter B. No difference in joint awareness after TKA: a matched-pair analysis of a classic implant and its evolutional design. Knee Surg Sports Traumatol Arthrosc. 2019 Jul;27(7):2124-2129. doi: 10.1007/s00167-019-05407-4. Epub 2019 Feb 14. PMID 30767068
- [Background] Behrend H, Hochreiter B, Potocnik P, El Baz Y, Zdravkovic V, Tomazi T. No difference in radiolucent lines after TKA: a matched-pair analysis of the classic implant and its evolutional design. Knee Surg Sports Traumatol Arthrosc. 2020 Dec;28(12):3962-3968. doi: 10.1007/s00167-020-05894-w. Epub 2020 Feb 15. PMID 32062683
- [Background] Bruggenjurgen B, Muehlendyck C, Gador LV, Katzer A. Length of stay after introduction of a new total knee arthroplasty (TKA)-results of a German retrospective database analysis. Med Devices (Auckl). 2019 Aug 7;12:245-251. doi: 10.2147/MDER.S191529. eCollection 2019. PMID 31496839
- [Background] Keogh CJ, Mulcahy D, Reidy D, Beverland DE, Harty JA. Polyethylene spinout in the Attune(R) Cruciate-Retaining Rotating-Platform (CR RP) total knee arthroplasty performed with a cruciate-sacrificing and measured-resection technique. Knee Surg Relat Res. 2020 Jul 22;32(1):36. doi: 10.1186/s43019-020-00057-0. PMID 32698908
- [Background] Giaretta S, Berti M, Micheloni GM, Ceccato A, Marangoni F, Momoli A. Early experience with the ATTUNE Total Knee Replacement System. Acta Biomed. 2019 Oct 29;90(12-S):98-103. doi: 10.23750/abm.v90i12-S.8997. PMID 31821292
- [Background] List R, Schutz P, Angst M, Ellenberger L, Datwyler K, Ferguson SJ; Writing Committee. Videofluoroscopic Evaluation of the Influence of a Gradually Reducing Femoral Radius on Joint Kinematics During Daily Activities in Total Knee Arthroplasty. J Arthroplasty. 2020 Oct;35(10):3010-3030. doi: 10.1016/j.arth.2020.05.039. Epub 2020 May 27. PMID 32564968
- [Background] Wiik AV, Aqil A, Tankard S, Amis AA, Cobb JP. Downhill walking gait pattern discriminates between types of knee arthroplasty: improved physiological knee functionality in UKA versus TKA. Knee Surg Sports Traumatol Arthrosc. 2015 Jun;23(6):1748-55. doi: 10.1007/s00167-014-3240-x. Epub 2014 Aug 27. PMID 25160471
- [Background] Beard DJ, Davies LJ, Cook JA, MacLennan G, Price A, Kent S, Hudson J, Carr A, Leal J, Campbell H, Fitzpatrick R, Arden N, Murray D, Campbell MK; TOPKAT Study Group. The clinical and cost-effectiveness of total versus partial knee replacement in patients with medial compartment osteoarthritis (TOPKAT): 5-year outcomes of a randomised controlled trial. Lancet. 2019 Aug 31;394(10200):746-756. doi: 10.1016/S0140-6736(19)31281-4. Epub 2019 Jul 17. PMID 31326135
- [Background] Stoddard JE, Deehan DJ, Bull AM, McCaskie AW, Amis AA. The kinematics and stability of single-radius versus multi-radius femoral components related to mid-range instability after TKA. J Orthop Res. 2013 Jan;31(1):53-8. doi: 10.1002/jor.22170. Epub 2012 Jun 13. PMID 22696446
- [Background] Dawson J, Fitzpatrick R, Murray D, Carr A. Questionnaire on the perceptions of patients about total knee replacement. J Bone Joint Surg Br. 1998 Jan;80(1):63-9. doi: 10.1302/0301-620x.80b1.7859. PMID 9460955
- [Background] Scott CEH, MacDonald DJ, Howie CR. 'Worse than death' and waiting for a joint arthroplasty. Bone Joint J. 2019 Aug;101-B(8):941-950. doi: 10.1302/0301-620X.101B8.BJJ-2019-0116.R1. PMID 31362549
- [Background] Behrend H, Giesinger K, Giesinger JM, Kuster MS. The "forgotten joint" as the ultimate goal in joint arthroplasty: validation of a new patient-reported outcome measure. J Arthroplasty. 2012 Mar;27(3):430-436.e1. doi: 10.1016/j.arth.2011.06.035. Epub 2011 Oct 13. PMID 22000572
- [Background] Feller JA, Bartlett RJ, Lang DM. Patellar resurfacing versus retention in total knee arthroplasty. J Bone Joint Surg Br. 1996 Mar;78(2):226-8. PMID 8666630
- [Background] Robinson RO, Herzog W, Nigg BM. Use of force platform variables to quantify the effects of chiropractic manipulation on gait symmetry. J Manipulative Physiol Ther. 1987 Aug;10(4):172-6. PMID 2958572
- [Background] O'Rourke MR, Callaghan JJ, Goetz DD, Sullivan PM, Johnston RC. Osteolysis associated with a cemented modular posterior-cruciate-substituting total knee design : five to eight-year follow-up. J Bone Joint Surg Am. 2002 Aug;84(8):1362-71. doi: 10.2106/00004623-200208000-00011. PMID 12177266
- See also: National Joint Registry for England, Wales, Northern Ireland and the Isle of Man, 17th Annual Report. (2020). Table 3.25 (a). — https://reports.njrcentre.org.uk/Portals/0/PDFdownloads/NJR%2017th%20Annual%20Report%202020.pdf
- See also: Australian Orthopaedic Association National Joint Replacement Registry Annual Report. (2020). Tables KT7. — https://aoanjrr.sahmri.com/documents/10180/689619/Hip%2C+Knee+%26+Shoulder+Arthroplasty+New/6a07a3b8-8767-06cf-9069-d165dc9baca7
- See also: Funk DA, Bridgens J. Confidence in the ATTUNE Knee is Driven by Real World Scientific Evidence: Response to Bonutti, et al. Article. (2017). — https://www.thieme-connect.com/products/ejournals/abstract/10.1055/s-0037-1608945
- See also: Stryker. Triathlon Total Knee System. — https://www.stryker.com/us/en/joint-replacement/products/triathlon-total-knee-system.html
- See also: Clary, C. Attune Knee System: Stability in Total Knee Replacement. DePuy Synthes Joint Reconstruction. — https://www.semanticscholar.org/paper/ATTUNE-TM-Knee-System-%3A-Stability-in-Total-Knee-Clary/7dc8c9144abc348b040147c500c8d0b7a2ccd96e